CLINICAL TRIAL: NCT07340502
Title: TACE Versus HAIC, Combined With PD-1 Inhibitors and Lenvatinib for Unresectable Hepatocellular Carcinoma: a Multicenter, Prospective, Observational Cohort Study
Brief Title: TACE Versus HAIC, Combined With PD-1 Inhibitors and Lenvatinib for Unresectable Hepatocellular Carcinoma
Status: Not yet recruiting | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Wan-Guang Zhang, Professor, Tongji Hospital
Other Study IDs: CHALLENGE-06
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: HCC
MeSH Terms: interventions — lenvatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TACE-based combination treatment cohort: Patients in this group were treated with TACE plus a PD-1 inhibitor and lenvatinib
  Interventions: Procedure: TACE; Drug: PD-1inhibitors; Drug: Lenvatinib
- HAIC-based combination treatment cohort: Patients in this group were treated with HAIC plus a PD-1 inhibitor and lenvatinib
  Interventions: Procedure: HAIC; Drug: PD-1inhibitors; Drug: Lenvatinib

INTERVENTIONS:
Procedure: TACE — TACE blocks the tumor's blood supply while delivering high concentrations of chemotherapy agents directly into the hepatic artery. Patients received on-demand TACE until the end of the study or tumor progression.
  Groups: TACE-based combination treatment cohort
Procedure: HAIC — HAIC involves the continuous infusion of high-dose chemotherapy into the hepatic artery via an indwelling catheter, enabling prolonged and deep tumor exposure. Patients received on-demand HAIC until the end of the study or tumor progression.
  Groups: HAIC-based combination treatment cohort
Drug: PD-1inhibitors — 200mg was given intravenously every three weeks.
Drug: Lenvatinib — The dose is determined by body weight, body weight greater than or equal to 60kg, 12mg, oral; Less than 60kg, 8mg, orally.

SUMMARY:
Although the combination of transarterial chemoembolization (TACE) with PD-1 inhibitor plus lenvatinib has become a new standard, the therapeutic efficacy for unresectable hepatocellular carcinoma (uHCC) still requires improvement, as TACE remains limited for patients with multifocal lesions, hypovascular tumors, or those complicated with portal vein tumor thrombosis (PVTT). Hepatic arterial infusion chemotherapy (HAIC), as an alternative locoregional therapy, has demonstrated advantages in treating these refractory cases. Therefore, this study innovatively designs a prospective cohort study to conduct a comparison of the two triple-combination regimens-"HAIC plus PD-1 inhibitor and lenvatinib" versus "TACE plus PD-1 inhibitor and lenvatinib"-in terms of real-world efficacy and safety, with a focus on enrolling patients who are likely to have suboptimal responses to TACE. This research aims to provide high-level evidence for selecting the optimal combined locoregional strategy for uHCC patients, thereby directly guiding clinical practice and potentially advancing the optimization of treatment strategies and personalized precision medicine to improve patient survival outcomes.

DETAILED DESCRIPTION:
This is a multicenter, prospective, observational cohort study designed to compare the efficacy and safety of transarterial chemoembolization (TACE) versus hepatic arterial infusion chemotherapy (HAIC), each combined with a programmed cell death protein-1 (PD-1) inhibitor and lenvatinib, for the treatment of unresectable hepatocellular carcinoma (uHCC), with a primary focus on progression-free survival (PFS). A total of 364 patients are planned to be enrolled and prospectively followed for efficacy and adverse events. The primary endpoint is PFS. Secondary endpoints include the objective response rate (ORR), overall survival (OS), and safety. Tumor response will be evaluated according to the modified Response Evaluation Criteria in Solid Tumors (mRECIST v1.1). Assessments will be performed every 56 days (with a ±3-day window) from the initiation of study treatment until disease progression, patient death, withdrawal of consent, loss to follow-up, or study termination (whichever occurs first). For patients who experience disease progression or initiate other antitumor therapies, survival follow-up will be conducted every 8 weeks (56 days, with a ±7-day window) from the time the event is documented to collect information on subsequent antitumor treatments and survival status until death, withdrawal of consent, loss to follow-up, or study termination.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 75 years;
* Tumor stage classified as BCLC-A to -C, with no evidence of extrahepatic metastasis;
* Newly diagnosed, treatment-naïve hepatocellular carcinoma with no prior anticancer therapy;
* Child-Pugh liver function score ≤ 7;
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1;
* Absence of severe organic diseases affecting major organs (e.g., heart, lung, brain).

Exclusion Criteria:

* Decompensated liver cirrhosis;
* Concurrent other malignancies or recurrent hepatocellular carcinoma;
* Any active, known, or suspected autoimmune disease;
* History of hypersensitivity to any component of PD-1 inhibitors or lenvatinib;
* Human immunodeficiency virus (HIV) infection; or active viral hepatitis (e.g., hepatitis B or C);
* Tumor thrombus involving the inferior vena cava, hepatic veins, or the main portal vein trunk.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a multicenter, prospective, observational cohort study designed to evaluate the efficacy and safety, primarily in terms of progression-free survival (PFS), of transarterial chemoembolization (TACE) versus hepatic arterial infusion chemotherapy (HAIC), each combined with a PD-1 inhibitor and lenvatinib, in the treatment of unresectable hepatocellular carcinoma (HCC). The study plans to enroll a total of 364 patients, who will be prospectively followed for treatment efficacy and adverse events. The primary endpoint is PFS. Secondary endpoints include the objective response rate (ORR), overall survival (OS), and safety.
Sampling Method: Probability Sample
Enrollment: 364 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From the date of enrollment, until the tumor progresses, the patient dies, or the study concludes (whichever occurs first), the assessment period can last up to 60 months.
  PFS was defined as the time from enrollment to tumor progression.

SECONDARY OUTCOMES:
Overall survival(OS) | From date of enrollment until the date of death from any cause, assessed up to 96 months.
  OS was defined as the time from enrollment to death.
Objective Response Rate (ORR) | From the date of enrollment, until the tumor progresses, the patient dies, or the study concludes (whichever occurs first), the assessment period can last up to 60 months.
  Objective Response Rate (ORR) is defined as the proportion of patients who achieve a best response of either complete response (CR) or partial response (PR) during a specified treatment period.

OTHER OUTCOMES:
Prespecified subgroup analyses | From the date of enrollment, until the patient dies, or the study concludes (whichever occurs first), the assessment period can last up to 60 months.
  Prespecified subgroup analyses were defined based on: (1) tumor distribution (confined to one hepatic lobe vs. involvement of both lobes); (2) tumor number (single vs. 2-3 vs. ≥3 tumors); and (3) tumor stage (BCLC stage A vs. B vs. C).

CONTACTS AND LOCATIONS:
Overall Officials: Wanguang Zhang, Principal Investigator — Tongji Hospital